CLINICAL TRIAL: NCT00073671
Title: Prevention of Depression in At-Risk Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Judith Garber, Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01MH064735 (NIH); R01MH064735 (NIH); DSIR 84-CTP (Other: NIH); R01MH064503 (NIH); R01MH064541 (NIH); R01MH064717 (NIH)
Record Dates: First submitted 2003-12-02; First posted 2003-12-03 (Estimated); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Depression
Keywords: Adolescent
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor were unaware of condition assignment
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1= Cognitive behavioral prevention of depression program (Experimental): Participants receive a group cognitive-behavioral prevention program, which involved 8 weekly sessions and 6 monthly sessions of CBT skills such as cognitive restructuring, problem-solving, assertivenss, and behavioral activation. Participants in this arm also were able to seek the same kinds of nonstudy treatments as described in the usual care arm.
  Interventions: Behavioral: Cognitive-behavioral prevention program
- 2 = Usual care (Active Comparator): Participants receive usual care, which involves any type of treatment (e.g., psychotherapy, counseling, pharmacotherapy).
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Cognitive-behavioral prevention program — Cognitive-behavioral prevention program includes 8 weekly and 6 monthly group sessions.
  Arms: 1= Cognitive behavioral prevention of depression program
Other: Usual care — Participants receive usual care
  Arms: 2 = Usual care

SUMMARY:
This study examines the impact of a group cognitive behavioral program aimed at preventing depressive disorders and symptoms in adolescents at risk for developing depression.

DETAILED DESCRIPTION:
Depression is a prevalent, chronic, and impairing condition that is often undetected and becomes more difficult to treat as chronicity increases. There is an increasing need to conduct large-scale depression prevention studies in adolescents. This study evaluates a cognitive-behavioral prevention (CBP) program to determine its effectiveness in preventing depressive disorders in at-risk adolescents. The study also will ascertain the costs this intervention to inform attempts at future dissemination of the program in "real world" settings.

Participants in this study are randomly assigned to receive either CBP for eight weekly and 6 monthly continuation sessions or usual care. Depressive symptoms and disorders, levels of functioning, and medical and mental health care utilization are assessed at baseline and again at 2, 8, 20, and 32 months after intake.

ELIGIBILITY:
Inclusion Criteria:

* A parent has had a depressive disorder during child's life
* Adolescent has had a past depressive episode or has current subsyndromal depressive symptoms measured on the Center for Epidemiological Studies Depression Scale (CES-D)

Exclusion Criteria:

* adolescent or parent ever diagnosed with bipolar I or schizophrenia;
* adolescent has a current DSM-IV mood disorder diagnosis

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 316 (Actual)
Dates: Start 2003-03; Primary Completion 2006-03 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Onset of a probable or definite depressive episodes (i.e., Depression Symptom Rating greater or equal to 4) | Time to a score of 4 or higher between baseline and 9 months using survival analysis
  a score of 4 or greater is considered an onset

SECONDARY OUTCOMES:
Number of depression-free days | Measured continuously through Month 33
  Using the depression symptom ratings (DSR) (1-6), each week is given a score of 1 to 6; depression-free days are those with ratings of 1 or 2 on the DSR.

CONTACTS AND LOCATIONS:
Overall Officials: Judy Garber, PhD, Principal Investigator — Vanderbilt University
Locations (4):
- United States (4):
  - Harvard University Medical School, Boston, Massachusetts
  - Kaiser Permanente Center for Health Research, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee

REFERENCES:
- [Result] Garber J, Clarke GN, Weersing VR, Beardslee WR, Brent DA, Gladstone TR, DeBar LL, Lynch FL, D'Angelo E, Hollon SD, Shamseddeen W, Iyengar S. Prevention of depression in at-risk adolescents: a randomized controlled trial. JAMA. 2009 Jun 3;301(21):2215-24. doi: 10.1001/jama.2009.788. PMID 19491183
- [Result] Beardslee WR, Brent DA, Weersing VR, Clarke GN, Porta G, Hollon SD, Gladstone TR, Gallop R, Lynch FL, Iyengar S, DeBar L, Garber J. Prevention of depression in at-risk adolescents: longer-term effects. JAMA Psychiatry. 2013 Nov;70(11):1161-70. doi: 10.1001/jamapsychiatry.2013.295. PMID 24005242
- [Result] Brent DA, Brunwasser SM, Hollon SD, Weersing VR, Clarke GN, Dickerson JF, Beardslee WR, Gladstone TR, Porta G, Lynch FL, Iyengar S, Garber J. Effect of a Cognitive-Behavioral Prevention Program on Depression 6 Years After Implementation Among At-Risk Adolescents: A Randomized Clinical Trial. JAMA Psychiatry. 2015 Nov;72(11):1110-8. doi: 10.1001/jamapsychiatry.2015.1559. PMID 26421861
- [Derived] Lynch FL, Dickerson JF, Clarke GN, Beardslee WR, Weersing VR, Gladstone TRG, Porta G, Brent DA, Mark TL, DeBar LL, Hollon SD, Garber J. Cost-Effectiveness of Preventing Depression Among At-Risk Youths: Postintervention and 2-Year Follow-Up. Psychiatr Serv. 2019 Apr 1;70(4):279-286. doi: 10.1176/appi.ps.201800144. Epub 2019 Jan 3. PMID 30929618
- [Derived] Weersing VR, Shamseddeen W, Garber J, Hollon SD, Clarke GN, Beardslee WR, Gladstone TR, Lynch FL, Porta G, Iyengar S, Brent DA. Prevention of Depression in At-Risk Adolescents: Predictors and Moderators of Acute Effects. J Am Acad Child Adolesc Psychiatry. 2016 Mar;55(3):219-26. doi: 10.1016/j.jaac.2015.12.015. Epub 2016 Jan 18. PMID 26903255